CLINICAL TRIAL: NCT04544761
Title: Resilience in People Following Spinal Cord Injury
Brief Title: Resilience in Persons Following Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Kiwanis Neurological Research Foundation (Unknown)
Responsible Party: Principal Investigator, Elliot Roth, Co-Medical Director, Brain Innovation Center, Shirley Ryan AbilityLab
Other Study IDs: STU00213014
Record Dates: First submitted 2020-09-04; First posted 2020-09-10 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Spinal Cord Injuries
Keywords: Resilience
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1-5 Years post: Persons with Spinal Cord Injury occurring between 1-5 years prior
  Interventions: Other: Structured Interview
- 5-15 Years post: Persons with Spinal Cord Injury occurring between 5-15 years prior
  Interventions: Other: Structured Interview
- >15 Years post: Persons with Spinal Cord Injury occurring at least 15 years prior
  Interventions: Other: Structured Interview

INTERVENTIONS:
Other: Structured Interview — Structured interview with research staff about your experience living with spinal cord injury

SUMMARY:
This study aims to quantify resilience in survivors of a spinal cord injury. The study will consist of structured interviews and self-reported surveys. We will look for common themes between participants at different stages of injury (1-5 years, 5-15 years, >15 Years).

DETAILED DESCRIPTION:
The goal of this project is to broaden the understanding of the lived experience of aging with a disability, from the perspectives of individuals with physical disabilities resulting from spinal cord injury (SCI). The specific objectives of this project are to:

1. Learn how people with SCI attain and maintain optimal quality of life as they age.
2. Understand how people with SCI develop resilience as they grow older.
3. Understand how individual quality of life is related to the degree and mechanism of resilience among people with SCI.
4. Learn which resources and practices have been most helpful and useful to people with SCI as they age with their disability.
5. Assess personal, behavioral, and environmental factors that contribute to resilience and quality of life among people aging with SCI.
6. Refine and confirm a holistic model for the relationships among the concepts of resilience, quality of life, and person-centered factors (resources, behaviors).

Through in-depth interviews and detailed surveys, we will explore how people with SCI attain and maintain optimal quality of life as they age, and how their quality of life relates to resiliency as they traverse the path of aging with SCI. We will explore with participants the resources and practices that have been most helpful and useful to them as they age with their disability.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* History of Traumatic Spinal Cord Injury at least 1 year prior
* Ability to self-report on factors affecting health and well being Exclusion Criteria
* Progressive Spinal Cord Injury

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons who have experienced spinal cord injury at least 1 year prior to enrollment
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Themes Survey | 1 day (Single time point)
  Common themes from the structured interviews

SECONDARY OUTCOMES:
Resilience | 1 day (Single time point)
  Measure of resilience from Connor-Davidson Resilience Scale [0-40], low score indicates greater resilience

OTHER OUTCOMES:
Health Questionnaire Surveys | 1 day (Single time point)
  Short Form-12 Health Survey [30-70] 50 indicates US average, values higher than 50 indicate better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Roth, MD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roth EJ, Lovell L, Barry A. Perspectives on factors influencing quality of life in persons with long-term spinal cord injury: a qualitative study. Spinal Cord. 2024 Jun;62(6):343-347. doi: 10.1038/s41393-024-00991-w. Epub 2024 Apr 22. PMID 38649756